CLINICAL TRIAL: NCT04594785
Title: Evaluation of Post Infectious Inflammatory Reaction (PIIR) in a Retrospective Study Concerning Children After Streptococcus Pneumoniae, Streptococcus Pyogenes and Neisseria Meningococcus Invasive Infection
Brief Title: Evaluation of Post Infectious Inflammatory Reaction (PIIR) Concerning Children After Streptococcus Pneumoniae, Streptococcus Pyogenes and Neisseria Meningococcus Invasive Infection
Acronym: RIPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0550
Record Dates: First submitted 2020-10-13; First posted 2020-10-20 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Streptococcus Pneumonia; Streptococcus Pyogenes Infection; Neisseria Meningitides Meningitis
Keywords: post-infectious inflammatory reactions; Neisseria Meningitis
MeSH Terms: conditions — Pneumonia; Streptococcal Infections; Meningitis, Meningococcal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As Covid 19 manifestations that have been recently described, inflammatory manifestation have major impact in infectious disease lesions. Some of them are delayed and provide Post infectious inflammatory reaction (PIIR), they are challenging for diagnosis and for management. Clinician have to avoid unnecessary antibiotic thearapy and in if necessary have to give immunosuppressive therapy. Except for rheumatic disease for group A streptococcus (GAS) infections there are not stanrdized diagnostic criteria and therapeutic protocol, and PIIR have probably a suboptimal management. In this context the investigators aim to explore PIIR in the 3 most frequent bacterial invasive infection in France, by a retrospective monocentric study. The investigators include all children betwwen 2012 and 2018 hospitalized for infections by Streptococcus pneumoniae (SP), Neisseria meningitidis (NM), and GAS invasive infections.

ELIGIBILITY:
Inclusion criteria:

* Less than 18 years of age
* Fever associated with GAS, NM, or SP invasive infection

Exclusion criteria:

* age > 18 years
* Impossibility to obtain the consent of parents / legal representatives.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Describe the frequency PIIRs | 1 day
  Describe the frequency PIIRs following invasive pneumococcal, meningococcal, or group A Streptococcal infection

SECONDARY OUTCOMES:
Characteristics PIIRs following invasive pneumococcal, meningococcal, or group A Streptococcal infection | 1 day
  Describe the characteristics PIIRs following invasive pneumococcal, meningococcal, or group A Streptococcal infection

OTHER OUTCOMES:
Predictors of PIIRs | 1 day
  Identified the predictors of PIIRs in order to find warning symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Eric JEZIORSKI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC